CLINICAL TRIAL: NCT00698139
Title: Cardiovascular and Neurohormonal Effects of Faster Atrial Pacing Rate for Six Hours in Patients With Congestive Heart Failure, Heart Rate <70 Beats Per Minute and Fluid Overload.
Brief Title: Cardiovascular and Neurohormonal Effects of Faster Atrial Pacing Rate
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed by Sponsor
Sponsor: Columbia University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Paolo Colombo, Herbert Irving Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAC6786
Record Dates: First submitted 2008-06-11; First posted 2008-06-17 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2014-07

CONDITIONS: Heart Failure
Keywords: heart failure; chronotropic incompetence
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention first, then control (Active Comparator): Ambulatory out-patients will be identified at Columbia-Presbyterian and New York University Medical Centers.
  On the first encounter, patients will come to clinic in the morning for baseline measurements. Subsequently, the atrial pacing rate will be increased to 85bpm for 6 hours. Patients will eat a standard breakfast provided by the hospital prior to the treatment session, and then will fast for the six-hour observation period. Patients will remain in supine position and will be clinically monitored for 6 hours. All patients will be on continuous cardiac monitors. Vital signs and symptoms of congestion/ischemia will be recorded every hour.
  On the second encounter, patients will come to clinic in the morning for baseline measurements.Subsequently, they will be given the illusion that their pacer has been adjusted, but the settings will remain unchanged. The rest of the protocol will be as described for the first encounter.
  Interventions: Device: Medtronic Pacemaker
- Control first, then intervention (Active Comparator): Ambulatory out-patients will be identified at Columbia-Presbyterian and New York University Medical Centers.
  On the first encounter, patients will come to clinic in the morning for baseline measurements.Subsequently, the control group will be given the illusion that their pacer has been adjusted, but the settings will remain unchanged. Patients will eat a standard breakfast provided by the hospital prior to the treatment session, and then will fast for the six-hour observation period. Patients will remain in supine position and will be clinically monitored for 6 hours. All patients will be on continuous cardiac monitors. Vital signs and symptoms of congestion/ischemia will be recorded every hour.
  On the second encounter, patients will come to clinic in the morning for baseline measurements. Subsequently, the atrial pacing rate will be increased to 85bpm for 6 hours. The rest of the protocol will be as described for the first encounter.
  Interventions: Device: Medtronic Pacemaker
- Intervention Only (Active Comparator): Ambulatory out-patients will be identified at Columbia-Presbyterian and New York University Medical Centers.
  Patients will come to clinic in the morning for baseline measurements. Subsequently, the atrial pacing rate will be increased to 85bpm for 6 hours. Patients will eat a standard breakfast provided by the hospital prior to the treatment session, and then will fast for the six-hour observation period. Patients will remain in supine position and will be clinically monitored for 6 hours. All patients will be on continuous cardiac monitors. Vital signs and symptoms of congestion/ischemia will be recorded every hour.
  Interventions: Device: Medtronic Pacemaker

INTERVENTIONS:
Device: Medtronic Pacemaker — Patients will come to clinic in the morning for baseline measurements. Subsequently, the atrial pacing rate will be increased to 85bpm for 6 hours. The control group will be given the illusion that their pacer has been adjusted, but the settings will remain unchanged. Patients will eat a standard breakfast provided by the hospital prior to the treatment session, and then will fast for the six-hour observation period. Patients will remain in supine position and will be clinically monitored for 6 hours. All patients will be on continuous cardiac monitors. Vital signs and symptoms of congestion/ischemia will be recorded every hour.
  Other Names: Medtronic Cardiac Resynchronization Therapy (CRT); Dual Chamber Pacemaker

SUMMARY:
Many patients with heart failure are unable to increase their heart rate appropriately when their body needs increased blood flow. As a result, they may be unable to mobilize excess fluid that their body retains. We hypothesize that we can provide assistance to their body in mobilizing this fluid by artificially increasing their heart rate using a pacemaker. We plan to conduct a prospective clinical trial to evaluate this hypothesis.

We will use a cross over design to study patients who already have biventricular pacemakers implanted or a narrow QRS and volume overload. We will screen them using a blood test that is a rough estimate of volume overload. Patients who meet the inclusion criteria will be randomly assigned to have their pacemakers adjusted or to have no intervention during the first of 2 visits. They will be unaware of which group they are in. Following adjustment, they will be monitored for six hours.

Prior to the pacemaker adjustment, several tests will be performed to evaluate heart function and the levels of hormones related that are affected by heart failure. These tests will be repeated at the end of the six hour intervention period in each visit. At the end of the visit patients who had their pacemakers adjusted will have it reset to their original settings.

DETAILED DESCRIPTION:
Many patients with heart failure suffer from chronotropic incompetence, an inability to raise their heart rate in response to metabolic demand. Previous studies have shown that brief increases in pacing rates in patients with biventricular pacemakers can improve cardiac contractility. We hypothesize that the benefits of an increased biventricular pacing rate could be sustained and would improve cardiovascular and neurohormonal parameters in patients suffering from volume overload. We intend to prospectively evaluate this hypothesis in a single blind randomized cross-over design trial.

We will screen 40 patients who have previously implanted biventricular pacemakers (or a narrow QRS) and an elevated B-type Natriuretic Peptide (BNP) level. Following enrollment, patients will be randomly assigned to have their atrial pacing rate increased to 85 beats per minute or to be unchanged during the first of 2 visits. Patients will be unaware of their treatment assignment. They will be observed for six hours in a monitored setting. The primary outcome will be cardiac output, as measured noninvasively by NICOM (Cheetah Medical Inc., Israel) system before and after the observation period. Secondary outcomes will include changes in neurohormonal measures and thoracic impedance. If this proof-of-concept study demonstrates a positive effect, future research would evaluate the ability of increased pacing rates to prevent or abort decompensation of Congestive Heart Failure (CHF).

ELIGIBILITY:
Inclusion Criteria:

1. Age>18
2. Congestive Heart Failure (CHF) (>6 months duration)
3. Left Ventricular Ejection Fraction (LVEF) <40%
4. Functional Class II-III
5. Stable oral treatment (>1 month),
6. Implanted Medtronic pacemaker/defibrillator with a) an atrial pacing lead and biventricular leads, or b) an atrial pacing lead and a single ventricular lead in patients with a narrow (normal) QRS complex (<120 msec) thus with no clinical indication for biventricular pacing.
7. Low heart rate (HR) (sinus rhythm (SR) or atrial pacing <70 bpm)
8. Symptomatically stable (with no clinical requirement for adjustments in medical therapy, i.e. diuretics)
9. Increase in intrathoracic fluid as evidenced by rain natriuretic peptide (BNP) >200.

Exclusion criteria:

1. Atrial fibrillation
2. Stable or unstable angina
3. Myocardial infarction within 6 months before the study
4. Intravenous inotropic support
5. Pregnant or breast feeding women. Women of child bearing potential must have a negative serum pregnancy test prior to enrollment.
6. Severe renal failure (creatinine> 2.5 mg/dl, hemodyalisis or peritoneal dialysis)
7. Known hepatic impairment (total bilirubin >3 mg/dL, albumin <2.8 mg/dL, or increased ammonia levels if performed)
8. Hemoglobin (hgb) <8 mg %, or active bleeding requiring transfusion

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Colombo, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall 3 subjects completed the study.
  One subject underwent the intervention only (i.e., 6 hours of faster pacing). Subsequently the protocol was modified to a prospective, randomized single-blind, cross over design. Two subjects completed the protocol according to this modification and underwent both real and sham intervention.
Period: Overall Study
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only
Started | 1 | 1 | 1
2nd Visit | 1 | 1 | 0 (1 subject in the Intervention Group did not have a 2nd visit (per design).)
Completed | 1 | 1 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only | Total
Number analyzed (Participants) | 1 | 1 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (0) | 85 (0) | 84 (0) | 69 (27)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 0 | 1
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Output (CO)
Description: The difference between post and pre CO
Time Frame: baseline and 6 hours
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only
Number analyzed (Participants) | 1 | 1 | 1
L/min
  1st Visit | -0.14 (0) | -0.05 (0) | 1.36 (0)
  2nd Visit | 0.95 (0) | 2.15 (0) | NA (NA) — Subject did not have a 2nd visit.

2. Secondary Outcome: Changes in Thoracic Impedence
Description: Impedence will be measured using the pacemaker programmer to determine the difference in thoracic impedence pre- and post-procedure.
Time Frame: baseline and 6 hours
Measure: Mean (Standard Deviation); unit: ohm
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only
Number analyzed (Participants) | 1 | 1 | 1
ohm
  1st Visit | 3.8 (0) | 0 (0) | 1.2 (0)
  2nd Visit | 2.6 (0) | -1.4 (0) | NA (NA) — Subject did not have a 2nd visit.

3. Secondary Outcome: Changes in B-type Natriuretic Peptide (BNP)
Description: B-type natriuretic peptide (BNP) was measured for all subjects to determint the difference between pre- and post-procedure.
Time Frame: baseline and 6 hours
Measure: Mean (Standard Deviation); unit: ng/L
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only
Number analyzed (Participants) | 1 | 1 | 1
ng/L
  1st Visit | 265 (0) | 19 (0) | 110 (0)
  2nd Visit | 261 (0) | 92 (0) | NA (NA) — Subject did not have a 2nd visit.

ADVERSE EVENTS:
Time Frame: 1 week
Description: telephone contact
Arm/Group | Intervention First, Then Control | Control First, Then Intervention | Intervention Only
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No